CLINICAL TRIAL: NCT02365324
Title: PAWS CLUB: Peer Education About Weight Steadiness
Brief Title: Peer Education About Weight Steadiness
Acronym: PAWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UIllinoisUC; 2012-68001-19652 (Other Grant/Funding Number: USDA National Institute of Food and Agriculture)
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2016-11

CONDITIONS: Obesity; Physical Activity
Keywords: culinary skills; menu planning; grocery shopping; children; healthy eating; physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-education Family Fitness Program (Experimental): Peer educators (children in grade 8) recruited from the schools participating in the study will be trained and will then be implementing the 12 week Peer-education Family Fitness Program (PE-FFP) intervention to children in 6th and 7th grade.
  Interventions: Behavioral: Peer-Education Family Fitness Program (PE-FFP)
- Family Fitness Program (FFP) (Other): Adult educators recruited from the University of Illinois Extension or the community will be trained and will then be implementing the 12 week Family Fitness Program (FFP) intervention to children in 6th and 7th grade.
  Interventions: Behavioral: Family Fitness Program (FFP)

INTERVENTIONS:
Behavioral: Peer-Education Family Fitness Program (PE-FFP) — The proposed integrated project will be implemented by peers and will evaluate the effects of an evidence-based extension education program, grounded in Stages of Change Learning Theory and guided by Social Cognitive Theory (SCT), having 2 arms for the study (with and without a peer-education mode of delivery) on balancing calories to manage body weight (BW), reducing certain foods and food components, increasing selected foods and nutrients, building healthy eating patterns [i.e., fundamental principles of the Dietary Guidelines for Americans (DGAs), 2010] and SCT variables.
  Other Names: PAWS Club: Peer-education About Weight Steadiness
  Arms: Peer-education Family Fitness Program
Behavioral: Family Fitness Program (FFP) — The proposed integrated project will be implemented by adults and will evaluate the effects of an evidence-based extension education program, grounded in Stages of Change Learning Theory and guided by Social Cognitive Theory (SCT), having 2 arms for the study (with and without a peer-education mode of delivery) on balancing calories to manage body weight (BW), reducing certain foods and food components, increasing selected foods and nutrients, building healthy eating patterns [i.e., fundamental principles of the Dietary Guidelines for Americans (DGAs), 2010] and SCT variables.
  Other Names: PAWS Club: Peer-education About Weight Steadiness
  Arms: Family Fitness Program (FFP)

SUMMARY:
The proposed integrated project will evaluate the effects of an evidence-based extension education program, Family Fitness Program (FFP) grounded in Stages of Change Learning Theory and guided by Social Cognitive Theory (SCT), with and without a peer-education mode of delivery on balancing calories to manage body weight (BW), reducing certain foods and food components, increasing selected foods and nutrients, building healthy eating patterns [i.e., fundamental principles of the Dietary Guidelines for Americans (DGAs), 2010] and SCT variables. Briefly, the 12-week program will target early adolescent children, ages 11-14 years, test a peer-education approach to behavioral change and will be delivered as an after-school program in local middle schools in support of childhood obesity prevention. Data will be collected at baseline (preintervention), after the 12-week program (post-intervention) and 6 months after completion of the program (maintenance).

DETAILED DESCRIPTION:
The 12-week intervention, either Family Fitness Program, FFP (adult-led control group) or Peer-education Family Fitness Program, PE-FFP (peer-led experimental group) will be delivered four times in each of the three schools participating in the study from May, 2015 to May 2017 as an after-school program to early adolescent children, ages 11-14 years, to partially meet the stated objectives in research. The proposed integrated project will follow a group-randomized controlled trial design. The intervention will be offered as an after-school programs in each of 3 schools (Urbana Middle School, Franklin Middle School and Mahomet Seymour-Junior High School). Programs will be conducted on Mondays, Tuesdays, Wednesday, and Thursdays for 12 weeks. After children are enrolled in the program, weekday by school will be randomly assigned to the adult-led FFP (control group) or to the peer-led PE-FFP (experimental group). This process will allow children the convenience of participating in the program on the day that is most compatible with their schedules, offer the control and experimental conditions at each of 2 schools and maintain randomization to treatment. Thus, each school will have 1 control group and 1 experimental group each time the program is conducted. Group randomization will occur during the fall-winter 2016 term and spring-summer 2017 term again. Data will be collected at baseline (pre-intervention), after the 12-week FFP or PE-FFP (post-intervention) and 6 months after completion of the program (maintenance). The FFP addresses all major elements of the Dietary guidelines for Americans (DGAs), 2010. Each weekly lesson will include: 1) 20-30 minutes of moderate physical activity; 2) nutrition activities; 3) discussions; 4) self-reflections; 5) goal setting activities for healthier eating and physical activity; 6) food and beverage tasting experiences; and 7) parent-child reflections. Lesson details are provided below. Incentive items will be distributed throughout the 12-week intervention. Adult educators will lead FFP lessons, while peer-educators will lead PE-FFP lessons. Study personnel will be present at each lesson, along with Illinois-Trans-disciplinary Obesity Prevention Program (I-TOPP) trainees to monitor each session and to conduct extension measures.

Lesson details:

1. Introduction to Fitness; For children: Introductions; ice-breakers; health and wellness; family physical activities and foods Energy balance; physical activity environment; body image; vegetables and fruits; family fitness For parents: An Introduction to family Fitness
2. Culinary Skills; For children: Knife safety; knife selection; cooking methods and utensils; focus on vegetables and fruits
3. Culinary Skills in Action; For children: Slicing, measuring, tasting vegetables and fruits; vegetable and fruit dishes
4. Physical Activity: Using Dietary Guidelines for Healthy Food Choices; For children and parents: Balancing calories to manage weight; energy; growth and development; growth charts; family physical activity values; building healthy eating patterns; nutrient-dense foods; flexible food patterns; vegetables and fruits; whole grains; seafood; family food choices; family food values
5. Breakfast for All; For children and parents: Increasing specific foods and nutrients; whole grains; vegetables and fruits; nutrients of concern (dietary fiber and potassium); flexible food patterns; family eating patterns; finding family time for healthy food choices and physical activities
6. Healthy Snacking and Healthy Food Choices; For children: Reducing certain foods and food components; energy-dense foods; solid fats and added sugars; sodium; refined grains; label reading (Nutrition Facts label); goal setting for food and snack choices; family snack choices For parents: Identifying and Overcoming Resistance to Change
7. Eating Out and Fast Foods; For children: Reducing certain foods and food components; label reading; menu reading; finding fats and oils; portion sizes; food advertising; food environment; eating at home with family or eating out choices
8. Healthy Beverages; For children: Increasing specific foods and nutrients; non-fat milk and dairy; water; nutrients of concern (calcium and vitamin D); food and health connections; practicing culinary skills
9. Setting Limits on Sweets and Fats; For children: Reducing certain foods and food components; finding fats and sugars in foods; practicing culinary skills; goal setting for food choices
10. Maintaining Physical Activity and Healthy Eating Patterns; For children: Balancing calories to maintain weight; Building healthy eating patterns; flexible approaches to eating; variety, balance and moderation; label reading; vegetables and fruits; whole grains; non-fat milk and dairy; seafood; oils; physical activities for the family
11. Family Menu Planning; Family food preferences and health needs; food costs and budgeting; family menus; shopping lists; family food purchasing
12. Grocery Shopping; For children: Field trip; in-store choices and selections; food costing; Wrap-Up

ELIGIBILITY:
Inclusion Criteria:

* Children in grade 6 or grade 7, 11-14 years old and their parents, enrolled in the schools participating in the study

Exclusion Criteria:

* Children younger than 11 years or older than 14 years, not enrolled in the schools participating in the study

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Demographic data | Evaluation at three time points: 0 months, 2 months and 8 months
  Children will complete a standardized questionnaire to provide age, gender, race/ethnicity, grade level and home address. Information about health (any acute or chronic illnesses) and health care services utilization (frequency of doctor's visits, use of specialists, medication use or need) will be provided by parents.
Goal setting tool | Evaluation at three time points: 0 months, 2 months and 8 months
  Children and parents will complete the Goal Setting for Family Fitness tool. Children and adults, respectively, will complete the Child or Adult versions of the Pre-Survey (baseline), Post-Survey (post-intervention) and Follow-Up Survey (6-months post-intervention).
Changes in 24-hour dietary intake recall | Evaluation at three time points: 0 months, 2 months and 8 months
  24-hour dietary intake recall completed by the multiple-pass method in an interview format.
Changes in 3-day dietary intake record | Evaluation at three time points: 0 months, 2 months and 8 months
  3-day dietary intake record (2 weekdays+1 weekend day).
Changes in 24-hour physical activity recall | Evaluation at three time points: 0 months, 2 months and 8 months
  Average energy expenditure of children (kcals/day) will be estimated from 1, 24-hour physical activity recall completed in an interview format.
Changes in 3-day physical activity record | Evaluation at three time points: 0 months, 2 months and 8 months
  3-day physical activity record (2 weekdays+1 weekend day).
Changes in Anthropometric measurements | Evaluation at three time points: 0 months, 2 months and 8 months
  In a private room with the child's parent present, a graduate research assistant (GRA) will measure the child's BW (kg) on a calibrated scale (Seca 700, Hanover, MD) to the nearest 0.1 kg and body height (cm) to the nearest 0.1 cm with a calibrated, standing stadiometer (Seca 700).
Changes in Social Cognitive Theory (SCT) variables | Evaluation at three time points: 0 months, 2 months and 8 months
  Social/family support, self-efficacy, self-regulation and outcome expectations for balancing calories to manage BW, reducing certain foods and food components, increasing selected foods and nutrients and building healthy eating patterns will be assessed by questionnaires.
Changes in blood pressure (BP) measurements | Evaluation at three time points: 0 months, 2 months and 8 months
  Seated systolic and diastolic BP (mmHg) will be measured by a trained GRA, using a sphygmomanometer (Baumanometer® Desk Model, Copiague, NY). Two BP measurements will be recorded with a 3-minute rest period between readings; values will be averaged.

SECONDARY OUTCOMES:
Process measure questionnaire | One questionnaire for each of the 12 sessions of the program (An average of six to twelve weeks)
  Program staff will administer the process measure questionnaire at the end of each session (12 sessions) to record information about participant attendance (children and adults), engagement during each weekly lessons and completion of program worksheets, and evaluate adult-educator and peer-educator program fidelity for each session for all control (FFP) and experimental (PE-FFP) groups.
Education measures | Once, at the end of the 12 week intervention
  The RE-AIM framework will be used as the foundation for measuring education and extension outcomes. Reach, efficacy, adoption, implementation and maintenance (REAIM) will be measured.
Extension measures | Once, at the end of the 12 week intervention
  Reach, Efficacy, Adoption, Implementation and Maintenance of the program will be determined at the end of the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nickols-Richardson, PhD, RD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (4):
- United States (4):
  - Franklin Middle School, Champaign, Illinois
  - Jefferson Middle School, Champaign, Illinois
  - Mahomet Seymour-Junior High School, Mahomet, Illinois
  - Urbana Middle School, Urbana, Illinois

REFERENCES:
- [Derived] Muzaffar H, Nikolaus CJ, Ogolsky BG, Lane A, Liguori C, Nickols-Richardson SM. Promoting Cooking, Nutrition, and Physical Activity in Afterschool Settings. Am J Health Behav. 2019 Nov 1;43(6):1050-1063. doi: 10.5993/AJHB.43.6.4. PMID 31662165